CLINICAL TRIAL: NCT07091162
Title: EValuation Of poLygenic Scores and CT imAging In Risk Factor Modification in Patients With diabEtes
Acronym: VOLTAIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Stephen Nicholls, Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VOLTAIRE-1
Record Dates: First submitted 2025-06-18; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. CTCA group (Active Comparator): Participants receive baseline CTCA results, in addition to standard care
  Interventions: Other: CTCA results
- 2. PRS group (Active Comparator): Participants receive polygenic risk score result, in addition to standard care
  Interventions: Other: PRS results
- 3. Control group (No Intervention): Participants receive standard care only with no additional information

INTERVENTIONS:
Other: CTCA results — Participants who are assigned to CTCA group will receive their CTCA results
  Arms: 1. CTCA group
Other: PRS results — Participants who are assigned to PRS group will receive their PRS results
  Arms: 2. PRS group

SUMMARY:
This study is a three-arm, parallel-group, randomised controlled trial evaluating the effect of using cardiac CT imaging or polygenic risk score in cardiovascular risk factor modification in patients with diabetes.

DETAILED DESCRIPTION:
The contemporary management of type 2 diabetes (T2D) involves a multifaceted model of care integrating intensive management of lipids, blood pressure, and glucose, along with lifestyle modifications. Despite these efforts, cardiovascular disease (CVD) remains a leading cause of morbidity and mortality among patients with T2D, largely due to suboptimal adherence to preventive strategies. The VOLTAIRE trial aims to assess the impact of providing personalised cardiovascular risk information derived from computed tomography coronary angiography (CTCA) and a polygenic risk score (PRS) on cardiovascular risk factor modification.

VOLTAIRE evaluates whether integrating CTCA and PRS into risk counselling enhances adherence to lifestyle and pharmacological interventions, ultimately improving cardiovascular outcomes among patients with T2D.

VOLTAIRE is a prospective three-arm, parallel-group, randomised controlled trial aiming to enrol 90 participants aged 40 years or older with T2D and no established atherosclerotic CVD. Participants will be randomised 1:1:1 to receive: (1) risk factor counselling plus CTCA result, (2) risk factor counselling plus PRS result or (3) standard risk factor counselling (control). Nurse-led motivational interviewing will be used for risk counselling. The primary outcome is change in non-calcified plaque volume measured by serial CTCA at 12 months. Secondary outcomes include low-density lipoprotein cholesterol levels, adherence to medication, patient engagement, CVD knowledge improvements, and psychological outcomes over 12 months.

VOLTAIRE seeks to determine if coupling nurse-led risk factor counselling with personalised CTCA or PRS information improves cardiovascular outcomes, adherence, and participant engagement in T2D management.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Established diagnosis of T2DM
* Having acceptable imaging quality as deemed by the VHI-AICL
* Able to have a PRS calculated

Exclusion Criteria:

* Unable to provide written informed consent.
* Unwilling to be followed for serial evaluation
* Clinically manifest CV disease
* Evidence of clinically significant coronary disease on CT that would preclude masking from participant's treating clinician for the duration of the study on the grounds of safety, including but not limited to, equal/greater than 50% in the left main coronary artery or equal/greater than 70% in any epicardial coronary artery
* Unable to participate in the study or complete protocol required assessments in the opinion of the Investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in non-calcified plaque volume, with Bonferroni correction at 12 months | From baseline CT to the end of study at 12 months

SECONDARY OUTCOMES:
Number of Participants achieving LDL-C <1.8 mmol/L | 12 months
Number of Participants who undergo intensification of lipid-lowering therapy | 12 months
  Intensification of lipid-lowering therapy at 12 months will be defined as the occurrence of any of the following:
  * an increase in the intensity of statin prescribed,
  * addition of ezetimibe, or
  * addition of a PCSK9 inhibitor (PCSK9i).
  This outcome will be assessed based on medication records at the 12-month follow-up.
Number of participants reporting high levels of adherence to their prescribed medications | 12 months
  Medication adherence will be assessed using a participant-reported item from a modified VOILS questionnaire at the 12-month follow-up. Participants are asked:
  "In the last week, I took my tablet(s):" with response options:
  * Every day
  * Almost every day
  * Less than half
  * Rarely or not at all
  Adherence will be defined as selecting "Every day", and the number of participants meeting this criterion will be reported.
Change in level of patient activation and engagement in their care, measured by PAM-13 questionnaire | 12 months
  Patient activation and engagement in care will be assessed using the 13-item Patient Activation Measure (PAM-13) at baseline and 12 months. Each item is scored on a 4-point Likert scale (Disagree Strongly to Agree Strongly), with responses converted into a continuous score ranging from 0 to 100.
  Higher scores indicate greater activation, reflecting better self-management and engagement in health care.
Change in depressive symptoms, measured by the Patient Health Questionnaire-9 (PHQ-9) | 12 months
  Depressive symptoms will be assessed using the 9-item Patient Health Questionnaire (PHQ-9). Each item is scored from 0 (not at all) to 3 (nearly every day), producing a total score from 0 to 27. Higher scores indicate more severe depressive symptoms. A higher score represents a worse outcome.
Change in anxiety symptoms, measured by the Generalized Anxiety Disorder-7 (GAD-7) scale | 12 months
  Anxiety will be assessed using the 7-item Generalized Anxiety Disorder scale (GAD-7). Each item is scored from 0 (not at all) to 3 (nearly every day), yielding a total score from 0 to 21. Higher scores indicate greater anxiety severity. A higher score represents a worse outcome.
Change in diabetes-related emotional distress, measured by the Diabetes Distress Scale (DDS-17) | 12 months
  Diabetes distress will be assessed using the 17-item Diabetes Distress Scale (DDS-17). Each item is scored on a 6-point Likert scale from 1 (not a problem) to 6 (a very serious problem). Mean item scores range from 1 to 6, with higher scores indicating greater distress. A higher score represents a worse outcome.
Change in health-related quality of life, measured by the EQ-5D-5L | 12 months
  Health-related quality of life will be assessed using the EQ-5D-5L questionnaire, which includes five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has five response levels, ranging from no problems to extreme problems. Responses will be converted into a health utility index score using the Australian-specific value set, ranging from <0 (worse than death) to 1 (perfect health). A higher utility score indicates better health status and quality of life.
Change in risk of obstructive sleep apnea, measured by the STOP-BANG questionnaire | 12 months
  Risk of obstructive sleep apnea will be assessed using the STOP-BANG questionnaire at baseline and 12 months. The tool includes 8 yes/no items: Snoring; Tiredness; Observed apnoea; High blood Pressure; Body mass index (BMI) >35 kg/m²; Age >50 years; Neck circumference >40 cm; Gender (male)
  Each "yes" is scored as 1 point, giving a total score from 0 to 8. Scores of: 0-2 = low risk; 3-4 = intermediate risk; 5-8 = high risk
  Higher scores indicate a higher risk of obstructive sleep apnea. Change in total STOP-BANG score will be reported.
Change in estimated 5-year cardiovascular disease (CVD) risk, measured by the NZSSD CVD Risk Calculator | 12 months
  Cardiovascular disease (CVD) risk will be assessed using the New Zealand Society for the Study of Diabetes (NZSSD) CVD Risk Assessment Calculator (www.nzssd.org.nz/cvd/). This tool estimates the 5-year absolute risk of a cardiovascular event based on patient characteristics, including age, sex, ethnicity, smoking status, diabetes status, blood pressure, lipids, and other clinical parameters.
  The calculator produces a score between 0% and >30%, with higher scores indicating greater risk.
Incidence of CVD events | 12 months
Number of participants achieving all three modifiable risk factor goals: LDL-C <1.8mmol/L, systolic blood pressure ≤130mmHg, and smoking cessation | 12 months
  This composite outcome reflects the number of participants who meet all of the following three modifiable risk factor goals at 12 months:
  * LDL-cholesterol < 1.8 mmol/L
  * Systolic blood pressure ≤ 130 mmHg
  * Smoking cessation (defined as self-reported non-smoking or validated by clinical records if available)
Change in hsCRP | 12 months
Change in HbA1c | 12 months
Change in total atheroma volume (TAV) measured by CTCA | 12 months
  Total atheroma volume (in mm³) will be assessed by CTCA at baseline and 12 months. TAV quantifies plaque burden in the coronary arteries. A higher TAV indicates more atherosclerotic plaque.
Change in calcified plaque volume measured by CTCA | 12 months
  Calcified plaque volume (in mm³) will be measured using CTCA at baseline and 12 months. It represents the volume of calcium-containing plaque within the coronary arteries. A higher volume indicates greater calcified atherosclerotic burden.
Change in pericoronary adipose tissue (PCAT) CT attenuation | 12 months
  PCAT attenuation will be measured in Hounsfield Units (HU) using CTCA. It reflects the inflammatory status of perivascular fat. Higher values are associated with greater coronary inflammation.

OTHER OUTCOMES:
Participant-reported appropriateness of the CTCA intervention | 12 months
  Appropriateness will be assessed using a custom participant survey and focus group interviews. Participants will rate whether they found the CTCA intervention relevant and suitable for their personal health needs. Responses will be summarised using Likert scales and thematic analysis.
Participant-reported feasibility of the CTCA intervention | 12 months
  Feasibility will be assessed through participant survey items and focus group discussions addressing clarity of instructions. Responses will be summarised using Likert scales and thematic analysis.
Participant-reported acceptability of the CTCA intervention | 12 months
  Acceptability will be measured using participant survey and focus group feedback on comfort, satisfaction, and willingness to undergo CTCA again. Ratings will be reported using Likert scales and thematic analysis.
Participant-reported appropriateness of the PRS intervention | 12 months
  Appropriateness will be assessed using a custom participant survey and focus group interviews. Participants will rate whether they found the PRS intervention relevant and suitable for their personal health needs. Responses will be summarised using Likert scales and thematic analysis.
Participant-reported feasibility of the PRS intervention | 12 months
  Feasibility will be assessed through participant survey items and focus group discussions addressing clarity of instructions. Responses will be summarised using Likert scales and thematic analysis.
Participant-reported acceptability of the PRS intervention | 12 months
  Acceptability will be measured using participant survey and focus group feedback on comfort, satisfaction, and willingness to undergo PRS testing again. Ratings will be reported using Likert scales and thematic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Nicholls, MBBS, PhD, Principal Investigator — Monash University
Locations (1):
- Victorian Heart Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
The Steering Committee will decide if and how IPD will be shared. It is expected that study Co Investigators will be able to access data once the primary results have been presented.